CLINICAL TRIAL: NCT06179030
Title: Systemic and Local Inflammatory Biomarkers in the Treatment of Refractory Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Büşra Çoban, Ophthalmology Resident, Saglik Bilimleri Universitesi
Other Study IDs: E-48670771
Record Dates: First submitted 2023-12-05; First posted 2023-12-21 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Macular Edema; Inflammation
Keywords: diabetic macular edema; biomarkers; inflammation; optical coherence tomography
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples (serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group 1: switched from bevacizumab to ranibizumab 0.5
  Interventions: Diagnostic Test: serum samples; Drug: dexamethasone implant versus ranibizumab
- Group 2: switched from bevacizumab to dexamethasone implant
  Interventions: Diagnostic Test: serum samples; Drug: dexamethasone implant versus ranibizumab

INTERVENTIONS:
Diagnostic Test: serum samples — The serum samples were taken from the patients at the 3rd month (switch point)
Drug: dexamethasone implant versus ranibizumab — dexamethasone implant versus ranibizumab will be studied as a secondary outcome

SUMMARY:
The current study aims to investigate the relationship between systemic inflammatory biomarkers and local inflammatory biomarkers on OCT in patients with treatment resistant diabetic macular edema(DME) and further explore the associations with treatment outcomes.

DETAILED DESCRIPTION:
This study was designed as a prospective open-label non rondomised observational study. The study was registered between April 18, 2022 and October 18, 2023. It is planned to include 80 volunteer patients over the age of 18 who are being followed up with the diagnosis of naive DME in the Retina Department of Prof Dr Cemil Tascioglu City Hospital and had poor response to the 3 consecutive initial monthly intravitreal bevacizumab loading dose. It was planned to evaluate systemic and local(OCT biomarker) inflammatory biomarker levels before swiching intravitreal agents, which may include intravitreal ranibizumab or intravitreal dexamethasone implant. The markers planned to be checked in blood samples are: IL-6, IL-8, TNF-a, ICAM-1, MCP-1, VEGF, HbA1c, CRP, ESR, haemogram, creatinine, AST, ALT, cholesterol. Patients were followed up monthly for 3 months after the switching. It was aimed to evaluate the level of systemic inflammatory biomarkers and the associations with treatment effectiveness. In addition, local OCT biomarkers (serous macular detachment and hyperreflective foci, etc.) and their relationship with treatment results were examined.

ELIGIBILITY:
Inclusion Criteria:

* who had refractory DME after 3 consecutive initial bevacizumab therapy
* treatment-naive

Exclusion Criteria:

* who had underwent anti-vegf treatment previously
* systemic inflammatory disease
* who had ocular surgery 6 months prior to enrollment
* uncontrolled hypertension
* <18 years old

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: treatment naive patients who were diagnosed with diabetic macular edema and had poor response to the 3 consecutive bevacizumab intravitreal injection loading phase.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
systemic inflammatory biomarkes correlates with OCT biomarkers and higher in poor responders | 6 months
  serum inflammatory biomarkers such as ICAM-1, MCP-1 , Il-6, IL-8, VEGF-A and TNFa will be studied. then, the levels of the aferometioned parameters will be compared with the treatment response and OCT parameters.

SECONDARY OUTCOMES:
The anatomical and visual recovery will be compared to dexamethasone versus ranibizumab | 6 months
  The groups will be compared regarding to anatomical and visual improvement. The anatomical improvement wil be assessed by central macular thickness measured by spectral domain OCT. The best corrected visual acuity change will be assessed by snellen and LogMAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided